CLINICAL TRIAL: NCT07297368
Title: Enhanced Tai Chi: A Randomised, Controlled, Single-Site Study of the Effects of Enhanced Tai Chi Training on Motor and Non-Motor Symptoms of Parkinson's Disease: A Pilot Study
Brief Title: Enhanced Tai Chi for Parkinson's Disease (Enhanced Tai Chi PD)
Acronym: ETC-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/WS/0099
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson's disease; Tai Chi; Enhanced Tai Chi; Qigong; Mind-body exercise; Non-pharmacological intervention; Balance training; Falls prevention; Motor symptoms; Non-motor symptoms; Quality of life; Pilot study; Feasibility study; Remote intervention; Hybrid trial
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 2:1 ratio to either the Enhanced Tai Chi intervention group (Enhanced-Tai-Chi-PD + usual treatment) or the control group (usual treatment only). The intervention group receives 36 sessions over 12 weeks (one in-person session and two remote sessions per week via Microsoft Teams). The control group continues with usual clinical care per local pathway. No crossover occurs between groups.
Who Masked: Outcomes Assessor
Masking Description: Baseline and Outcome assessments are performed by a blinded rater who is not involved in intervention delivery and does not have access to group allocation. Participants and care providers are not masked due to the nature of the behavioural intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Tai Chi + Usual Treatment (Experimental): Participants receive the Enhanced Tai Chi intervention in addition to usual clinical care. Enhanced Tai Chi consists of 36 structured one-hour sessions delivered over 12 weeks (three sessions per week: one in-person session and two remote sessions via Microsoft Teams). Participants are encouraged to undertake short additional home practice. Attendance is recorded to monitor adherence. Usual clinical care continues as directed by the treating physician.
  Interventions: Behavioral: Enhanced Tai Chi (Enhanced-Tai-Chi-PD)
- Usual Treatment (Control) (Active Comparator): Participants continue standard clinical care as determined by their treating physician (stable dopaminergic medications, and referrals to physiotherapy, occupational therapy, speech and language therapy as clinically needed). No Tai Chi is provided during the study period.
  Interventions: Other: Usual Treatment (Standard Clinical Care)

INTERVENTIONS:
Behavioral: Enhanced Tai Chi (Enhanced-Tai-Chi-PD) — Participants assigned to this arm receive Enhanced Tai Chi, a structured mind-body exercise program adapted specifically for people with Parkinson's disease. The program consists of 36 one-hour sessions delivered over 12 weeks (3 sessions/week: 1 in-person studio session and 2 remote sessions via Microsoft Teams). The intervention incorporates seven movement components including Qi Gong, single and double silk-reeling, standing energy/postural work, balance walking, Fa Jin (energy release), and a ten-direction balance form. Sessions focus on balance, postural control, fluid movement, coordination, breathing, and body alignment. Participants are encouraged to complete short additional home practice, and session attendance is logged to monitor compliance.
  Arms: Enhanced Tai Chi + Usual Treatment
Other: Usual Treatment (Standard Clinical Care) — Participants continue standard clinical care for Parkinson's disease as determined by their treating physician. No Enhanced Tai Chi or other study-specific exercise intervention is provided during the study period.
  Arms: Usual Treatment (Control)

SUMMARY:
This pilot study evaluates whether a structured, Parkinson's disease-specific Tai Chi programme ("Enhanced Tai Chi") can improve motor and non-motor symptoms in people with Parkinson's disease (PD).

PD is a progressive neurological condition associated with motor impairments such as bradykinesia, rigidity, gait disturbance and postural instability, as well as non-motor symptoms including fatigue, pain, mood disturbance, sleep problems and cognitive changes. Although pharmacological treatments improve many motor symptoms, balance and postural control often respond poorly, contributing to falls and reduced independence.

Enhanced Tai Chi is a tailored programme developed specifically for people with PD, incorporating elements of Tai Chi and Qi Gong focused on balance control, coordination, postural alignment, body awareness and confidence in movement. This single-site, randomised, controlled pilot trial will enrol 30 adults with idiopathic PD (Hoehn & Yahr stages I-III), randomised in a 2:1 ratio to Enhanced Tai Chi plus usual clinical care or usual clinical care alone.

Participants in the intervention group will complete 36 supervised one-hour sessions over 12 weeks (three sessions per week: one in-person and two delivered remotely), with optional independent practice encouraged. Adherence will be monitored through attendance records. Outcomes will be assessed at baseline, post-intervention and 3-month follow-up. Findings will inform feasibility, acceptability and preliminary efficacy estimates to support the design of a future definitive randomised controlled trial.

DETAILED DESCRIPTION:
Background and Rationale

Parkinson's disease (PD) is a progressive neurodegenerative disorder characterised by motor and non-motor symptoms that substantially affect quality of life and functional independence. While dopaminergic therapies remain the cornerstone of treatment, symptoms such as balance impairment and postural instability often respond incompletely, increasing the risk of falls and injury. Exercise-based interventions are increasingly recommended as adjunctive therapies in PD and may improve mobility, balance, non-motor symptoms and overall quality of life.

Tai Chi and related mind-body practices emphasise slow, controlled movements, weight shifting, postural control, breathing and mental focus. Previous studies suggest Tai Chi may improve balance and reduce falls in people with PD; however, many trials vary in methodological quality and provide limited detail regarding intervention content. Enhanced Tai Chi for Parkinson's (Enhanced-Tai-Chi-PD) was developed to address these limitations by providing a structured, PD-specific programme targeting balance, proprioception, coordination and movement confidence.

Study Design

This is a single-site, randomised, controlled, interventional pilot study. Thirty adults with idiopathic Parkinson's disease will be randomised in a 2:1 ratio to either Enhanced Tai Chi plus usual clinical care or usual clinical care alone. Assessments will be conducted at baseline, after completion of the 12-week intervention period, and at 3-month follow-up.

Intervention

Participants allocated to the intervention arm will attend three one-hour sessions per week for 12 weeks (36 sessions total), comprising one in-person session and two remotely delivered sessions via a secure video platform. The programme consists of seven structured movement components adapted for Parkinson's disease, including Qi Gong-based exercises, silk-reeling movements, balance walking, standing postural exercises and coordinated directional movement forms. Optional independent practice is encouraged. Attendance and adherence will be recorded throughout the intervention period.

Participants in the control arm will continue with usual clinical care as determined by their treating clinicians.

Safety, Data Handling and Oversight

Adverse events, serious adverse events and medication changes will be monitored throughout the study. Study data will be pseudonymised and stored securely in accordance with General Data Protection Regulation (GDPR) requirements and Good Clinical Practice. The study has received appropriate ethical and institutional approvals.

Expected Outcomes

This pilot trial will generate preliminary data on feasibility, adherence and effect size estimates for Enhanced Tai Chi in Parkinson's disease. Results will inform the design and power calculations of a future definitive randomised controlled trial evaluating this intervention as a scalable, low-risk adjunct to standard Parkinson's disease care.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (Hoehn & Yahr stage I-III)
* Able to stand and participate in movement sessions
* Stable medication dose for ≥ 4 weeks before study entry

Exclusion Criteria:

* Atypical or secondary parkinsonism
* Advanced therapies (DBS, apomorphine infusion, jejunal levodopa)
* Dementia (MoCA ≤ 21)
* Other neurological or medical conditions limiting participation
* Inability to commit to scheduled sessions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in motor symptoms (MDS-UPDRS Part III) | Baseline to 12 weeks (end of intervention)
  Clinician-rated assessment using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale, Part III (MDS-UPDRS III), performed in the ON medication state. Total score ranges from 0 to 132, with higher scores indicating greater motor impairment. Reductions in score indicate improvement in motor symptoms.

SECONDARY OUTCOMES:
Change in non-motor symptoms (MDS Non-Motor Symptoms Scale) | Baseline, 12 weeks, and 3-month follow-up
  Assesses frequency and severity of non-motor symptoms in Parkinson's disease. Total score ranges from 0 to 360, with higher scores indicating greater non-motor symptom burden. Interpretation of scores is as follows: Mild (1-44 points), Moderate (45-78 points), Severe (79-112 points), and very severe (>112).
Patient Global Impression of Change (PGIC) | 12 weeks and 3-month follow-up
  Participant-reported overall perception of change in health status. Scored on a 7-point Likert scale (1 = very much improved, 4 = no change, 7 = very much worse). Lower scores indicate perceived improvement, while higher scores indicate worsening.
Change in quality of life (PDQ-8) | Baseline, 12 weeks, and 3-month follow-up
  Self-reported measure of health-related quality of life. Total score ranges from 0 to 32, with lower scores indicating better quality of life. A decrease in score reflects improvement. For this study, a meaningful change is defined as a change of 5-7 points, indicating clinical significant impact to quality of life.
Change in cognitive function (MoCA) | Baseline, 12 weeks, and 3-month follow-up
  Brief cognitive screening tool. Total score ranges from 0 to 30, with higher scores indicating better cognitive function. Scores 26-30 (normal), 18-25 (mild cognitive impairment), 10-17 (moderate cognitive impairment), and <10 (severe cognitive impairment). Increases in score suggest improvement or preservation of cognitive function.
Change in pain (King's Parkinson's Disease Pain Scale - KPPS) | Baseline, 12 weeks, and 3-month follow-up
  Clinician-rated assessment of Parkinson's disease-related pain across multiple domains. Total score ranges from 0 to 168, with higher scores indicating greater pain severity. Lower scores represent improvement in pain symptoms. Interpretation for this study: score 0 (no pain), scores 17-34 (mild to moderate), 68-70 (moderate to severe). Minimal clinical important difference is measured by a change of 3 points to indicate meaningful change.
Change in sleep disturbance (PD Sleep Scale-2) | Baseline, 12 weeks, and 3-month follow-up
  Assesses sleep disturbances in Parkinson's disease. Total score ranges from 0 to 60, with higher scores indicating worse sleep quality. For this study, meaningful change is defined as a decrease of at least 3.44 points for improvement or an increase of at least 2.07 points for worsening.
Change in fatigue (Parkinson's Fatigue Scale-16) | Baseline, 12 weeks, 3-month follow-up
  Self-reported fatigue severity scale. Total score ranges from 16 to 80, with higher scores indicating greater fatigue.
Change in anxiety and depression (Hospital Anxiety and Depression Scale - HADS) | Baseline, 12 weeks, and 3-month follow-up
  Self-reported assessment of anxiety and depression using two subscales (HADS-A and HADS-D). Each subscale ranges from 0 to 21, with higher scores indicating greater symptom severity. Scores 0-7 (normal), 8-10 (mild/borderline), 11-14 (moderate), and 15-21 (severe). Lower scores indicate improvement in anxiety and/or depressive symptoms. Meaningful change is defined as change of 2 points.
Change in apathy (Apathy Scale - AS) | Baseline, 12 weeks, 3-month follow-up
  Self-reported measure of apathy. Total score ranges from 0 to 42, with higher scores indicating greater apathy. PD patients with scores over 14 suggest clinically significant meaningful apathy. Lower scores represent improvement in motivational symptoms.
Change in physical activity level (PASE) | Baseline, 12 weeks, 3-month follow-up
  Self-reported assessment of physical activity over the previous week. Scores typically range from 0 to >400, with higher scores indicating greater levels of physical activity. Increases in score indicate higher activity levels.
Change in global clinical severity (CISI-PD) | Baseline, 12 weeks, 3-month follow-up
  Clinician-rated global assessment across four domains (motor signs, disability, cognitive status, and complications). Each domain is scored from 0 to 6, giving a total score range of 0 to 24, with higher scores indicating greater disease severity. A reduction in total score over time indicates clinical improvement.
Change in balance performance (Berg Balance Scale) | Baseline, 12 weeks, 3-month follow-up
  Clinician-rated 14-item assessment of balance performance. Total score ranges from 0 to 56, with higher scores indicating better balance. For this study we consider 0-20 (wheelchair/ high fall risk), 21-40 (needing aids/ moderate risk), 41-56 (independent, low risk), with scores <45 indicating increased risk of falls for the PD population. Increases in score indicate improvement in balance ability.
Change in mobility (Timed Up and Go - TUG) | Baseline, 12 weeks, 3-month follow-up
  Performance-based assessment measuring the time (in seconds) required to stand from a seated position, walk 3 meters, turn, return, and sit down. Lower times indicate better mobility and functional performance. For this study with PD patients our scoring is as follows: <12 seconds (good mobility), 12-14 seconds (differentiates PD fallers vs non-fallers, with higher end being riskier), >14 seconds (high risk for fall), >20 seconds (needs assistance for basic transfer), and >30 seconds (limited mobility, decreased independence).
Change in walking speed (10-Meter Walk Test) | Baseline, 12 weeks, 3-month follow-up
  Performance-based assessment measuring the time (in seconds) to walk 10 meters at a comfortable pace. Lower times indicate faster walking speed and improved gait performance. For this study, there needs to be a minimum detectable change of approximately 0.18 m/s (comfortable) or 0.25 m/s (fast) to show real improvement, not just testing variation.
Number of monthly falls | Baseline, 12 weeks, 3-month follow-up
  Self-reported number of falls recorded using participant-maintained fall diaries. Higher values indicate increased fall frequency, while reductions indicate improvement in fall risk.
Feasibility / compliance with intervention | Continuous over 12-week intervention
  17a. Intervention adherence: Percentage of scheduled Enhanced Tai Chi sessions attended during the intervention period. Values range from 0% to 100%, with higher percentages indicating better adherence.
  17b. Intervention tolerability: Proportion of participants who discontinue the intervention due to tolerability issues. Values range from 0 to 100%, with lower percentages indicating better tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Whitney, MSc, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request after publication of primary results. Data access request can be made by contacting our Research Data team for the study (kch-tr.taichi.inbox@nhs.net)
Supporting Information: Study Protocol, SAP
Time Frame: Post publication of data (earliest 01-DEC-2026)